CLINICAL TRIAL: NCT07398183
Title: Effects of Digitally Delivered Parent-based Behavioural Sleep Intervention in Children With Autism Spectrum Disorder (ASD) - A Randomised Controlled Trial
Brief Title: Sleep Intervention in Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA240518
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Insomnia; Autism Spectrum Disorder (ASD)
Keywords: insomnia; Autism spectrum disorder; ASD; behavioral sleep intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App-based CBT-I with personalised telephone support (Experimental): App-based cognitive behavioural therapy for insomnia with personalised telephone support
  Interventions: Behavioral: App-based CBT-I with personalised telephone support
- App-based CBT-I without personalised support (Experimental): App-based cognitive behavioural therapy for insomnia without personalised telephone support
  Interventions: Behavioral: App-based CBT-I without personalised telephone support
- TAU group (No Intervention): Participants will continue their usual clinical follow-up and receive standard treatment where needed. No app-based intervention and telephone support will be provided to this group.

INTERVENTIONS:
Behavioral: App-based CBT-I with personalised telephone support — Participants in this group will be instructed to download a smartphone application. The smartphone app-based intervention, involving six sequential modules, is structured and based on the well-established behavioural sleep intervention elements for managing sleep problems in children, with the consideration of catering to the needs of children with ASD. The main treatment components include: (1) psychoeducation about sleep in the developmental context as well as in the context of ASD, (2) sleep hygiene education, (3) sleep-focused behavioural strategies (e.g., consistent bedtime routine, bedtime fading, extinction, sleep restriction, use of 'bedtime pass'), (4) relaxation strategies, (5) cognitive restructuring (targeting dysfunctional cognitions) and (6) relapse prevention. A weekly phone call support by a trained therapist, using a semi-structured script, will be provided during the intervention period (around 15 mins each time) to the parents.
  Other Names: App-based intervention with personalised support
  Arms: App-based CBT-I with personalised telephone support
Behavioral: App-based CBT-I without personalised telephone support — Participants in this group will be instructed to download the same smartphone application used in the app-based CBT-I with personalised support. No telephone support will be provided to this group.
  Other Names: App-based intervention without personalised support
  Arms: App-based CBT-I without personalised support

SUMMARY:
The goal of this randomised controlled trial is to examine the following research questions: 1) whether digitally delivered parent-based behavioural sleep intervention with or without personalised support is effective in improving sleep, clinical and daytime symptoms, and 2) whether such interventions can also improve parental sleep, mental health, and parenting stress in children with ASD and insomnia.

DETAILED DESCRIPTION:
A randomised, assessor-blind, parallel-group controlled trial (RCT) will be conducted in children with ASD and insomnia. Eligible participants will be randomised to one of the following groups: app-based cognitive behavioural therapy for insomnia (CBT-I) with personalised support, app-based CBT-I without personalised support, or treatment-as-usual (TAU). Randomisation will be carried out using an automated online system and stratified by gender. Assessments will be conducted at pre-treatment and post-treatment (1 week after intervention completion). The two active treatment groups will be additionally followed up at post-treatment 3 months and posttreatment 6 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) Parents/caregivers with a child aged 6 to 12 years old, and attending a local mainstream primary school at the time of recruitment;
* (2) The child is diagnosed to have ASD, which will be based on the assessment conducted by a psychiatrist or a clinical psychologist that incorporates the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) assessment criteria, with corroboration by the Autism Diagnostic Interview - Revised (ADI-R);
* (3) The child is reported by the parent/caregiver to have insomnia symptoms, typically a difficulty in falling asleep with or without bedtime resistance, which is operationally defined as sleep onset latency exceeding 25 minutes and occurring three or more times per week. The child's sleep problems have lasted for a minimum of three months and have led to an impairment in the daily functioning of the child and/or parents. Such inclusion criteria are based on the DSM-V criteria for insomnia, with the choice of a 25-minute sleep onset latency criteria based on the normative values reported by Scholle et al.;
* (4) Parent owns and knows how to use smartphones and can comprehend Chinese language;
* (5) The child's parent or guardian gives written informed consent of participation into the study;
* (6) Being able to comply with the study protocol.

Exclusion Criteria:

* (1) Children with diagnosed intellectual disability;
* (2) Children with any diagnosed co-morbid neurological or medical conditions which could have affected their sleep, such as blindness, traumatic brain injury, epilepsy and poorly controlled eczema;
* (3) Children with diagnosed sleep disorders other than insomnia or with suspected sleep apnoea (as assessed by the Children's Sleep Habits Questionnaire (CSHQ): obtaining a score of 4 or above on the sleep-disordered breathing subscale on the CSHQ) that may potentially contribute to a disruption in sleep continuity and quality. Children who are currently receiving regular melatonin treatment, as well as other medications such as Selective Serotonin Reuptake Inhibitors (SSRIs), will be considered for inclusion in the trial if they continue to meet the eligibility criteria.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Child: Change of child's sleep problems | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The Children's Sleep Habits Questionnaire (CSHQ) - parent report is a commonly used measure to assess sleep symptoms in children aged 4-12 years. It consists of 33 items to evaluate a child's sleep behavior over the past week. Items are rated on a 3-point scale to indicate the frequency of each sleep behavior: "usually/five to seven times per week," "sometimes/two to four times per week," and "rarely/zero to once per week." The CSHQ total score is the sum of the 33 questions and ranges from 33 to 99. Higher scores indicate more severe sleep disturbances.

SECONDARY OUTCOMES:
Child: Change of child's ASD symptoms | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The Social Communication Questionnaire, Current Form - parent report (SCQ-CF-PR) is a 40-item screening instrument designed to assess social communication deficits and repetitive behavioral patterns associated with autism spectrum disorder (ASD). This scale quantifies autistic characteristics aligned with the three core domains of impairment in ASD: communication, reciprocal social interaction, and restricted, repetitive, and stereotyped (RRS) behaviors. The SCQ-CF-PR yields a total raw score ranging from a minimum of 0 to a maximum of 40 points, with higher scores indicating greater severity of ASD-related social communication and behavioral impairments.
Child: Change of child's emotional and behavioural problems | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The Strengths and Difficulties Questionnaire (SDQ) - parent report is a 25-item instrument for measuring internalising and externalising problems in children and adolescents. It consists of five domains (emotional symptoms, conduct problems, hyperactivity/inattention, peer problems, and prosocial behaviours), with 5 items each rated on a three-point scale [0 ("not true") to 2 ("certainly true")]. The conduct problem and hyperactivity/inattention domains were grouped under the externalizing problem subscale (range 0-20), while the emotional symptoms and peer problems were grouped under the internalizing problem subscale (range 0-20). The total difficulties score is generated by summing the scores from the four problem scales (excluding Prosocial Behavior), yielding a range from 0 to 40. Higher scores indicate more problems, except that a higher prosocial score indicated better prosocial behaviours.
Child: Change of child's executive function | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) - Parent Report is a 63-item questionnaire designed to assess executive functioning deficits in children and adolescents across everyday home and community settings. The scale generates nine clinical subscale raw scores and a single Global Executive Composite (GEC) raw score (the primary summary measure of overall executive functioning). All raw scores range from a minimum of 0 to subscale/maximum-specific maximum values (total GEC raw score: 0-189). Higher raw scores indicate greater severity of executive functioning impairments.
Child: Change of child's daytime sleepiness | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Pediatric Daytime Sleepiness Scale (PDSS) - parent report is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Child: Change of child's quality of life | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The Pediatric Quality of Life Inventory 4.0 (PedsQL) - parent report is a validated 23-item measure of quality of life for children aged 2 to 18 years. Each item is rated on a 5-point Likert scale from "never" to "almost always" based on the behavior of child in the past month. The scores are transformed on a scale from 0 to 100, with a higher score indicating better quality of life.
Child: Change of parent-reported child sleep diary measures | Baseline, Post-Treatment (1 week after intervention completion) for all consented participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Parent-reported child's daily sleep diary for consecutive seven days. Sleep diary derived parameters include: 1) time in bed (TIB) in hours. 2) total sleep time (TST) in hours. 3) sleep onset latency (SOL) in mins. 4) wake after sleep onset (WASO) in mins. 5) sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %.
Child: Change of child's actigraphy-based measures | Baseline, Post-Treatment (1 week after intervention completion) for all consented participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for these participants in the treatment groups.
  The child's sleep-wake pattern will be objectively measured by 7-day wrist actigraphy. Sleep parameter estimated by actigraphy will include time in bed, total sleep time, sleep onset latency (SOL), wake after sleep onset (WASO), and sleep efficiency.
Child: Change of overall severity of child's clinical symptoms | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of psychopathology, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.
Parent: Change of parental insomnia symptoms | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Insomnia Severity Index (ISI) is a 5-item self-rated scale to measure insomnia symptoms. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.
Parent: Change of parental sleep quality | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Parent: Change of parental mental health | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Depression Anxiety Stress Scales-21 (DASS-21) consists of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS scales contains 7 items. Each subscale ranges from 0 to 21. Higher scores suggest more depression, anxiety and stress, respectively.
Parent: Change of parenting stress | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Parenting Stress Index-Short Form (PSI-SF) is a 36-item self-report measure designed to assess stress in the parent-child relationship, derived from the full Parenting Stress Index. It includes three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (PCDI), and Difficult Child (DC). Each subscale has 12 items rated on a 5-point Likert scale, amounting to a total score that ranges from 36 to 180. Higher scores indicate higher levels of stress in the parent-child relationship.
Parent: Change of parental quailty of life | Baseline, Post-Treatment (1 week after intervention completion) for all participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The World Health Organisation- Five Well-Being Index (WHO-5) consists of 5 self-report items designed to measure subjective well-being. Each item is rated on a 6-point scale from 0 ("at no time") to 5 ("all of the time"), resulting in a raw score range of 0 to 25. Higher scores indicate better well-being.
Parent: Change of parental sleep diary measures | Baseline, Post-Treatment (1 week after intervention completion) for all consented participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  Daily sleep diary for consecutive seven days. Sleep diary derived parameters include: 1) time in bed (TIB) in hours. 2) total sleep time (TST) in hours. 3) sleep onset latency (SOL) in mins. 4) wake after sleep onset (WASO) in mins. 5) sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %.
Parent: Change of parental actigraphy-based measures | Baseline, Post-Treatment (1 week after intervention completion) for all consented participants, and additionally two follow-ups at Post-Treatment 3-month and Post-Treatment 6-month for participants in the treatment groups.
  The parental sleep-wake pattern will be objectively measured by 7-day wrist actigraphy. Sleep parameter estimated by actigraphy will include time in bed, total sleep time, sleep onset latency (SOL), wake after sleep onset (WASO), and sleep efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong